CLINICAL TRIAL: NCT02264717
Title: Dan-NICAD - Danish Study of Non-Invasive Diagnostic Testing in Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Dan-NICAD
Record Dates: First submitted 2014-09-26; First posted 2014-10-15 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Angina Pectoris; Arteriosclerosis; Coronary Artery Disease; Myocardial Ischemia
MeSH Terms: conditions — Angina Pectoris; Arteriosclerosis; Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cardiac MRi (Active Comparator): A minimum of 150 patients will be randomized to Cardiac MRI followed by conventional angiography CCA-FFR, after detection of obstructive anatomic coronary artery stenoses on coronary Computed Tomography Angiography (cCTA)
  Interventions: Procedure: Cardiac MRI
- SPECT (Active Comparator): A minimum 150 patients will be randomized to SPECT followed by conventional angiography CCA-FFR, after detection of obstructive anatomic coronary artery stenoses on coronary Computed Tomography Angiography (cCTA).
  Interventions: Procedure: SPECT

INTERVENTIONS:
Procedure: SPECT — Patients are randomized to either SPECT or Cardiac MRI
  Arms: SPECT
Procedure: Cardiac MRI — Patients are randomized to either SPECT or Cardiac MR
  Arms: Cardiac MRi

SUMMARY:
1. The primary purpose of this study is to determine the diagnostic accuracy of the CADscore System, a new danish technology that records sounds from turbulence of bloodflow in the coronary vessels.

And secondary:

1. To determine the accuracy of cardiac magnetic resonance imaging (MRI) and single-photon emission computed tomography (SPECT), as secondary tests after detection of obstructive anatomic coronary artery stenosis by coronary computed tomographic angiography (CCTA).
2. To examine the patient population for bio-genetic markers related to development of arteriosclerosis.
3. To evaluate virtual fractional flow reserve (vFFR) computed from coronary angiograms.

DETAILED DESCRIPTION:
Primary study CCTA is currently the first choice to rule out coronary artery disease (CAD) in patients with typical or atypical chest pain. 4500 patients are annually examined with CCTA, in the Central Jutland Region of Denmark, and approximately 80% are discharged after ruling out CAD. CCTA is a diagnostic scan that exposes the patients to radiation, therefore a better risk stratification prior to the test is desirable. The CADscore is a newly developed danish technology that has been tested so far in 1000 patients. An area under the curve of the receiver operating characteristic (AUC of ROC) of 75-80 has been determined compared to conventional coronary angiography using quantitative coronary angiography (CCA-QCA). This indicates that the CADscore could potentially be used to diagnose CAD as a supplement or risk stratification prior to CCTA.

We aim to evaluate the CADscore in a large clinical trial including 2000 patients that by clinical indication undergo cCTA. After cCTA approximately 20 % (400 patients) will need evaluation by CCA with FFR. CADscore results will be compared to CCTA and CCA-QCA. Secondary, the CADscore will be compared to the results of CCA-FFR and perfusion scans, Cardiac-MRI and SPECT.

Substudies

1. Perfusion scans

   CCTA demonstrates good diagnostic performance for detection and exclusion of anatomic coronary artery stenosis, but several studies have previously shown that CCTA has a low positive predictive value for identification of hemodynamically significant CAD. This emphasizes the need for additional tests to evaluate the severity (or exclusion) of hemodynamically significant CAD. Measurement of FFR during CCA represents the "gold standard" for assessment of the hemodynamic significance of coronary artery stenosis. The disadvantage of CCA with FFR is that it is an invasive procedure.

   After cCTA approximately 20 % (400 patients) will need further testing and that group of patients will be randomized to either Cardiac MRI or SPECT followed by CCA with FFR.

   The substudy aims to evaluate the diagnostic accuracy of perfusion imaging (Cardiac MRI and SPECT) compared with CCA with FFR.
2. Virtual FFR

The accuracy and precision of virtual-FFR compared with conventional FFR will be determined. Virtual FFR is computed from the coronary angiogram using computational fluid dynamics. Subjects with diameter stenosis in the range of 30 to 90% by visual estimate in one or more vessel segments with reference diameter ≥2.0 mm will be included in the analysis. FFR is the reference standard to determine the presence or absence of hemodynamically significant obstruction with a cut-off value of 0.80. Computation of vFFR with and without hyperaemia will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Indication for Cardiac CT
* Signed

Exclusion Criteria:

* Age under 40
* Pregnant, potentially pregnant or breast feeding
* Contraindication for adenosine (severe asthma, clinical aortic stenosis)
* Reduced kidney function (eGFR < 40 ml/min)
* Contraindication for MRI
* Previous history of allergy to contrast
* Previous revascularisation procedure

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1676 (Actual)
Dates: Start 2014-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of the CADscore system compared to CCTA and CCA-QCA. | Within one week before or after CCTA
  Diagnostic precision will be evaluated as the AUC-ROC. The CADscore will be dichotomized at cut off values of 20,25 and 30 and performance reported with sensitivity, specificity, positive predictive value, negative predictive value and diagnostic accuracy. The CADscore system operates with 3 intervals of risk stratification: <20, 20-30, >30 (low, intermedia and high risk of cardio vascular disease, respectively) Obstructive CAD is defined as ≥ 50% diameter stenosis as determined by quantitative analysis of CCA (QCA). Non-Obstructive CAD is defined as no detection of obstructive anatomic coronary artery stenosis by CCTA or stenosis detected by CCTA combined with a evaluation by CCA-QCA demonstrating a luminal stenosis diameter < 50 %.

SECONDARY OUTCOMES:
Safety of CADScore Safety of CADScore | One week after the use of CADScore
  Registration of adverse events related to the use of CADScore
Diagnostic accuracy of the CADScore system compared to CCA-FFR. | Within four weeks after CADScore
  Diagnostic precision will be evaluated as the AUC-ROC and performance reported with sensitivity, specificity, positive predictive value, negative predictive value and diagnostic accuracy.
  CAD is defined as CCA-FFR under 0.80.

OTHER OUTCOMES:
Feasibility of virtual FFR | one day
  Feasibility of vFFR compared to conventional FFR assessed as fraction of conventional FFR measurements where a vFFR values is computed by the core lab.
Diagnostic accuracy of virtual FFR | one day
  Diagnostic accuracy of vFFR as the area under the receiver operating characteristic curve (AUC by ROC). The performance of vFFR in predicting functionally significant stenosis is assessed with and without hyperaemia using sensitivity, specificity, positive predictive value, negative predictive value and diagnostic accuracy, together with their 95% confidence intervals.
The diagnostic accuracy of perfusion imaging (Cardiac MRI and SPECT) | Within 4 weeks after the CCTA
  Diagnostic performance will be evaluated as the AUC-ROC, sensitivity, specificity, positive predictive value, negative predictive value and diagnostic accuracy.
  CAD is defined as a CCA-FFR below 0,80. A Chi2 test will be used to compare SPECT and Cardiac-MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Morten Bøttcher, MD, Ph.D, Principal Investigator — Regional Hospital of Herning, department of cardiology
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Aarhus, Central Jutland
  - Regional Hospital of Herning, Herning, Central Jutland
  - Regional Hospital of Silkeborg, Silkeborg, Central Jutland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Westra J, Rasmussen LD, Karim SR, Jensen RV, Ejlersen JA, Gormsen LC, Bottcher M, Eftekhari A, Winther S, Christiansen EH. Coronary microvascular disease in patients referred to coronary angiography following coronary computed tomography angiography. EuroIntervention. 2025 Sep 1;21(17):e1005-e1014. doi: 10.4244/EIJ-D-24-01155. PMID 40887988
- [Derived] Rasmussen LD, Sikjaer M, Soby JH, Pedersen OB, Westra J, Efthekhari A, Christiansen EH, Foldyna B, Williams MC, Dweck MR, Newby DE, Douglas PS, Bottcher M, Winther S. Dual probability approach for risk adjustment in patients with a low clinical likelihood of coronary artery disease. Eur Heart J Cardiovasc Imaging. 2025 Aug 29;26(9):1507-1517. doi: 10.1093/ehjci/jeaf193. PMID 40590244
- [Derived] Brix GS, Rasmussen LD, Rohde PD, Nissen L, Nyegaard M, O'Donoghue ML, Bottcher M, Winther S. Elevated lipoprotein(a) levels are independently associated with the presence of significant coronary stenosis in de-novo patients with stable chest pain. Am Heart J. 2025 Apr;282:103-113. doi: 10.1016/j.ahj.2025.01.001. Epub 2025 Jan 7. PMID 39788470
- [Derived] Pedersen G, Dahl JN, Rasmussen LD, Garm Blavnsfeldt AB, Bottcher SH, Bottcher MH, Nyegaard M, Nissen L, Winther S. Biomarkers for identification of high-risk coronary artery plaques in patients with suspected coronary artery disease. J Cardiovasc Comput Tomogr. 2024 Sep-Oct;18(5):467-475. doi: 10.1016/j.jcct.2024.06.009. Epub 2024 Jul 2. PMID 38955554
- [Derived] Moller PL, Rohde PD, Dahl JN, Rasmussen LD, Nissen L, Schmidt SE, McGilligan V, Gudbjartsson DF, Stefansson K, Holm H, Bentzon JF, Bottcher M, Winther S, Nyegaard M. Predicting the presence of coronary plaques featuring high-risk characteristics using polygenic risk scores and targeted proteomics in patients with suspected coronary artery disease. Genome Med. 2024 Mar 20;16(1):40. doi: 10.1186/s13073-024-01313-8. PMID 38509622
- [Derived] Moller PL, Rohde PD, Dahl JN, Rasmussen LD, Schmidt SE, Nissen L, McGilligan V, Bentzon JF, Gudbjartsson DF, Stefansson K, Holm H, Winther S, Bottcher M, Nyegaard M. Combining Polygenic and Proteomic Risk Scores With Clinical Risk Factors to Improve Performance for Diagnosing Absence of Coronary Artery Disease in Patients With de novo Chest Pain. Circ Genom Precis Med. 2023 Oct;16(5):442-451. doi: 10.1161/CIRCGEN.123.004053. Epub 2023 Sep 27. PMID 37753640
- [Derived] Westra J, Rasmussen LD, Eftekhari A, Winther S, Karim SR, Johansen JK, Hammid O, Sondergaard HM, Ejlersen JA, Gormsen LC, Mogensen LJH, Bottcher M, Holm NR, Christiansen EH. Coronary Artery Stenosis Evaluation by Angiography-Derived FFR: Validation by Positron Emission Tomography and Invasive Thermodilution. JACC Cardiovasc Imaging. 2023 Oct;16(10):1321-1331. doi: 10.1016/j.jcmg.2023.02.008. Epub 2023 Apr 12. PMID 37052562
- [Derived] Winther S, Nissen L, Schmidt SE, Westra J, Andersen IT, Nyegaard M, Madsen LH, Knudsen LL, Urbonaviciene G, Larsen BS, Struijk JJ, Frost L, Holm NR, Christiansen EH, Botker HE, Bottcher M. Advanced heart sound analysis as a new prognostic marker in stable coronary artery disease. Eur Heart J Digit Health. 2021 Mar 19;2(2):279-289. doi: 10.1093/ehjdh/ztab031. eCollection 2021 Jun. PMID 36712398
- [Derived] Christiansen MK, Winther S, Nissen L, Vilhjalmsson BJ, Frost L, Johansen JK, Moller PL, Schmidt SE, Westra J, Holm NR, Jensen HK, Christiansen EH, Guethbjartsson DF, Holm H, Stefansson K, Botker HE, Bottcher M, Nyegaard M. Polygenic Risk Score-Enhanced Risk Stratification of Coronary Artery Disease in Patients With Stable Chest Pain. Circ Genom Precis Med. 2021 Jun;14(3):e003298. doi: 10.1161/CIRCGEN.120.003298. Epub 2021 May 25. PMID 34032468
- [Derived] Therkildsen J, Nissen L, Jorgensen HS, Thygesen J, Ivarsen P, Frost L, Isaksen C, Langdahl BL, Hauge EM, Boettcher M, Winther S. Thoracic Bone Mineral Density Derived from Cardiac CT Is Associated with Greater Fracture Rate. Radiology. 2020 Sep;296(3):499-508. doi: 10.1148/radiol.2020192706. Epub 2020 Jul 14. PMID 32662758
- [Derived] Christiansen MK, Nissen L, Winther S, Moller PL, Frost L, Johansen JK, Jensen HK, Guethbjartsson D, Holm H, Stefansson K, Botker HE, Bottcher M, Nyegaard M. Genetic Risk of Coronary Artery Disease, Features of Atherosclerosis, and Coronary Plaque Burden. J Am Heart Assoc. 2020 Feb 4;9(3):e014795. doi: 10.1161/JAHA.119.014795. Epub 2020 Jan 25. PMID 31983321
- [Derived] Winther S, Nissen L, Westra J, Schmidt SE, Bouteldja N, Knudsen LL, Madsen LH, Frost L, Urbonaviciene G, Holm NR, Christiansen EH, Botker HE, Bottcher M. Pre-test probability prediction in patients with a low to intermediate probability of coronary artery disease: a prospective study with a fractional flow reserve endpoint. Eur Heart J Cardiovasc Imaging. 2019 Nov 1;20(11):1208-1218. doi: 10.1093/ehjci/jez058. PMID 31083725
- [Derived] Westra J, Tu S, Winther S, Nissen L, Vestergaard MB, Andersen BK, Holck EN, Fox Maule C, Johansen JK, Andreasen LN, Simonsen JK, Zhang Y, Kristensen SD, Maeng M, Kaltoft A, Terkelsen CJ, Krusell LR, Jakobsen L, Reiber JHC, Lassen JF, Bottcher M, Botker HE, Christiansen EH, Holm NR. Evaluation of Coronary Artery Stenosis by Quantitative Flow Ratio During Invasive Coronary Angiography: The WIFI II Study (Wire-Free Functional Imaging II). Circ Cardiovasc Imaging. 2018 Mar;11(3):e007107. doi: 10.1161/CIRCIMAGING.117.007107. PMID 29555835
- [Derived] Winther S, Nissen L, Schmidt SE, Westra JS, Rasmussen LD, Knudsen LL, Madsen LH, Kirk Johansen J, Larsen BS, Struijk JJ, Frost L, Holm NR, Christiansen EH, Botker HE, Bottcher M. Diagnostic performance of an acoustic-based system for coronary artery disease risk stratification. Heart. 2018 Jun;104(11):928-935. doi: 10.1136/heartjnl-2017-311944. Epub 2017 Nov 9. PMID 29122932
- [Derived] Nissen L, Winther S, Isaksen C, Ejlersen JA, Brix L, Urbonaviciene G, Frost L, Madsen LH, Knudsen LL, Schmidt SE, Holm NR, Maeng M, Nyegaard M, Botker HE, Bottcher M. Danish study of Non-Invasive testing in Coronary Artery Disease (Dan-NICAD): study protocol for a randomised controlled trial. Trials. 2016 May 26;17(1):262. doi: 10.1186/s13063-016-1388-z. PMID 27225018